CLINICAL TRIAL: NCT07334119
Title: A Phase 1, Open-Label, First-in-Human, Dose Escalation Study to Investigate the Safety, Pharmacokinetics, Pharmacodynamics and Preliminary Efficacy of MT-304 in Adults With Advanced HER2-Expressing Solid Tumors
Brief Title: Safety, Pharmacokinetics, Pharmacodynamics and Preliminary Efficacy of MT-304 in Adults With Advanced HER2-Expressing Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Myeloid Therapeutics (Industry)
Collaborators: CREATE Medicines (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MTX-HER2-304
Record Dates: First submitted 2025-11-14; First posted 2026-01-12 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-10

CONDITIONS: HER2-Expressing Solid Tumors
Keywords: Anti-HER2 chimeric antigen receptor; Chimeric Antigen Receptor (CAR); mRNA; Lipid nanoparticle (LNP); Urothelial carcinoma; Endometrial carcinoma; Ovarian epithelial carcinoma; Breast carcinoma (all subtypes); Gastric adenocarcinoma; Esophageal adenocarcinoma; Non-small cell lung cancer; Colorectal carcinoma; Biliary cancer (including Gallbladder carcinoma and extrahepatic cholangiocarcinoma)
MeSH Terms: conditions — Carcinoma, Transitional Cell; Endometrial Neoplasms; Carcinoma, Ovarian Epithelial; Breast Neoplasms; Adenocarcinoma Of Esophagus; Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms; Biliary Tract Neoplasms; Cholangiocarcinoma | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MT-304 Monotherapy (Experimental): Participants receive MT-304 administered intravenously once every 14 days (Q14D) in escalating dose levels.
  Interventions: Drug: MT-304
- MT-304 + Nivolumab Combination Therapy (Experimental): Participants receive MT-304 administered intravenously once every 14 days (Q14D) in combination with nivolumab as "per local label" administered once every 28 days (Q28D).
  Interventions: Drug: MT-304 + Nivolumab

INTERVENTIONS:
Drug: MT-304 — Safety, tolerability, and pharmacokinetics will be evaluated.
  Other Names: mRNA-LNP
  Arms: MT-304 Monotherapy
Drug: MT-304 + Nivolumab — Combination therapy begins after monotherapy dose clearance by the Safety Review Committee.
  Other Names: mRNA-LNP
  Arms: MT-304 + Nivolumab Combination Therapy

SUMMARY:
This clinical trial is designed to evaluate the safety, pharmacokinetics, pharmacodynamics, and preliminary efficacy of MT-304 in adults with advanced HER2-expressing solid tumors. The main questions it aims to answer are:

* What is the safety profile of MT-304 when administered alone or with nivolumab?
* What is the recommended Phase 2 dose (RP2D) of MT-304?

Participants will:

* Receive MT-304 alone (every 14 days) or with nivolumab (every 28 days).
* Attend regular clinic visits for assessments and monitoring.
* Continue treatment until disease progression, unacceptable toxicity, or study discontinuation.

DETAILED DESCRIPTION:
This multicenter, open-label, Phase 1 trial is designed to assess the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), and preliminary efficacy of MT-304 in adults aged 18 and older with advanced HER2-expressing solid tumors.

The study consists of two treatment modules:

* Module 1 (Monotherapy): Participants receive MT-304 every 14 days for 28-day cycles, with dosing adjustments based on clinical benefit and safety evaluations.
* Module 2 (Combination Therapy): Participants receive MT-304 in combination with nivolumab, administered every 14 days and 28 days, respectively, also allowing for dosing adjustments.

The Bayesian Optimal Interval (BOIN) design will guide dose escalation, overseen by a Safety Review Committee to establish the recommended Phase 2 dose (RP2D).

Regular assessments, including vital signs and laboratory tests, will monitor safety and efficacy throughout the trial, with follow-up visits for up to 2 years post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or above
* Histologically confirmed diagnosis of metastatic or advanced epithelial cancer expressing HER2 (Note: Participants with other tumor types expressing HER2 may be considered pending discussion with the Medical Monitor).
* Measurable lesion per RECIST 1.1 criteria.
* Eastern Cooperative Oncology Group (ECOG) performance status Grade of 0 or 1.
* Adequate Organ function

Exclusion Criteria:

* Known active CNS metastasis and/or carcinomatous meningitis.
* Any acute illness including fever.
* History of symptomatic congestive heart failure
* History of (noninfectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
* Uncontrolled pleural effusion, pericardial effusion, or ascites
* Active autoimmune disease not related to prior therapy for primary malignancy that has required systemic therapy in the last 1 year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-01-31 (Estimated); Study Completion 2028-03-30 (Estimated)

PRIMARY OUTCOMES:
Type, incidence and severity of Adverse Events | Up to 90 days from the last dose of Investigational Medicinal Product (IMP)
  Safety and tolerability profile assessed by the Common Terminology Criteria for Adverse Events v5.
Number of Participants With Change From Baseline in Vital Signs (Composite Safety Outcome) | Up to 30 days from the last dose of IMP
  Body temperature, body weight, pulse rate, and blood pressure (systolic and diastolic) assessed collectively; participants with clinically significant changes in any vital sign parameter will be summarized as a composite safety outcome.
Number of Participants With Abnormal Clinical Laboratory Parameters (Composite Safety Outcome) | Up to 30 days from the last dose of IMP
  Hematology, clinical chemistry, coagulation, virology testing, and urinalysis assessed collectively; participants with abnormalities in any laboratory parameter will be summarized as a composite safety outcome.
Number of Participants With Change From Baseline in ECG Parameters (Composite Safety Outcome) | Screening through Day 28, with assessments performed on Screening, Day 1 (pre-dose), and Day 28.
  PR interval, QRS duration, QT interval, corrected QT interval (QTc), and heart rate assessed collectively from 12-lead ECG recordings; participants with clinically significant changes in any ECG parameter will be summarized as a composite safety outcome.
Maximum Tolerated Dose (MTD) | 28 days from the last dose of IMP
  The MTD in Module 1 (monotherapy) will be determined based on dose-limiting toxicities (DLTs).
Optimal Biological Dose (OBD) | 28 days from the last dose of IMP
  The OBD in Module 2 (combination) will be identified based on dose-limiting toxicities (DLTs).

SECONDARY OUTCOMES:
Pharmacokinetics (PK) | From Day 1, Day 2, Day 8, and Day 15 of Cycles 1 and 2, and Day 1 of Cycle 3 (each cycle is 28 days).
  PK Parameter: Maximum plasma concentration (Cmax)
Pharmacokinetics (PK) | From Day 1, Day 2, Day 8, and Day 15 of Cycles 1 and 2, and Day 1 of Cycle 3 (each cycle is 28 days).
  PK parameter: Area under Curve
Pharmacokinetics (PK) | From Day 1, Day 2, Day 8, and Day 15 of Cycles 1 and 2, and Day 1 of Cycle 3 (each cycle is 28 days).
  PK parameter: Time of maximum observed plasma concentration (tmax)
Pharmacokinetics (PK) | From Day 1, Day 2, Day 8, and Day 15 of Cycles 1 and 2, and Day 1 of Cycle 3 (each cycle is 28 days).
  PK parameter:Terminal half-life (t½)
Pharmacokinetics (PK) | From Day 1, Day 2, Day 8, and Day 15 of Cycles 1 and 2, and Day 1 of Cycle 3 (each cycle is 28 days).
  PK parameter: Plasma Clearance (CL)
Pharmacokinetics (PK) | From Day 1, Day 2, Day 8, and Day 15 of Cycles 1 and 2, and Day 1 of Cycle 3 (each cycle is 28 days).
  PK parameter: Volume of Distribution (Vd)
Pharmacokinetics (PK) | From Day 1, Day 2, Day 8, and Day 15 of Cycles 1 and 2, and Day 1 of Cycle 3 (each cycle is 28 days).
  PK parameter: Mean residence time (MRT)
To assess adverse events of special interest (AESI) by measuring infusion reaction | Upto 90 days from the last dose of IMP
To assess adverse events of special interest (AESI) by measuring cytokine release syndrome (CRS) | Upto 90 days from the last dose of IMP
To assess adverse events of special interest (AESI) by measuring immune effector cell-associated neurotoxicity syndrome (ICANS) | Upto 90 days from the last dose of IMP
To assess adverse events of special interest (AESI) by measuring hypersensitivity reaction | Upto 90 days from the last dose of IMP
To assess the incidence of second primary malignancies reported as adverse events of special interest (AESI) occurring during the study treatment period and long-term follow-up. | From first dose of Investigational Medicinal Product (IMP) through end of study and follow-up (up to 2 years)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Maurer, MD, Study Director — Myeloid Therapeutics
Locations (3):
- Australia (3):
  - Calvary Mater Newcastle, Waratah, New South Wales
  - Scientia Clinical Research Ltd, Randwick, New South Wales (nsw)
  - Linear Clinical Research, Nedlands, Western Australia

IPD SHARING:
Plan to Share IPD: No